CLINICAL TRIAL: NCT02019563
Title: Mineral Trioxide Aggregate/Ferric Sulfate Pulpotomy for Vital Primary Incisors: A Randomized Controlled Trial
Brief Title: MTA/FS Pulpotomy for Vital Primary Incisors: A Randomized Controlled Trial
Acronym: MTA/FS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Peter Judd, Dentist-in-Chief, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000019443
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Dental Caries; Dental Pulp Exposure
Keywords: pediatrics; dental caries; dental pulp exposure; incisor
MeSH Terms: conditions — Dental Caries; Dental Pulp Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MTA/FS pulpotomy Group (Experimental): Children randomized to this arm will undergo a mineral trioxide aggregate (MTA) pulpotomy after hemostasis is achieved using ferric sulfate (FS).
  Interventions: Procedure: MTA/FS pulpotomy Group
- RCT Group (Active Comparator): Children randomized to this group will undergo the root canal therapy (RCT) technique.
  Interventions: Procedure: RCT Group

INTERVENTIONS:
Procedure: RCT Group — After complete removal of all caries, if a pulp exposure is detected the pulp chamber will be opened and the pulp tissue removed. The canal will be irrigated with water and then filled with non-reinforced ZOE.
  Arms: RCT Group
Procedure: MTA/FS pulpotomy Group — After complete removal of all caries, if a pulp exposure is detected the pulp chamber will be opened and vital coronal pulp to a depth of 2mm below free gingival margin will be removed. A solution of ferric sulfate will be applied to the amputated pulp surface and then flushed with water. MTA paste is then used to cover over the exposed amputated pulp surface.
  Arms: MTA/FS pulpotomy Group

SUMMARY:
To compare radiographic and clinical outcomes and survival of mineral trioxide aggregate/ferric sulfate (MTA/FS) pulpotomy and root canal therapy (RCT) in carious vital primary maxillary incisors.

DETAILED DESCRIPTION:
Dental caries is the most common chronic disease in children. Caries of the primary maxillary incisors is common in young children; often necessitating either extraction or pulp therapy. The premature loss of primary maxillary incisors can adversely affect a child's dental occlusion, ability to properly size food boluses for swallowing, speech articulation, facial esthetics and psychosocial development. Pulp treatment of cariously exposed vital primary incisors may prevent premature tooth loss as well as eliminate pain. Currently, there is a paucity of outcome investigations with regard to pulp therapy in primary incisors.

ELIGIBILITY:
Inclusion Criteria:

* children with one or more carious primary maxillary incisors where removal of dental caries will likely to produce a vital pulp exposure
* reside in the GTA at time of inclusion
* English-speaking

Exclusion Criteria:

* history of spontaneous or lingering stimulated pain, swelling, fistula or sinus tract, tenderness to percussion and pathological mobility
* incisors with preoperative radiographic evidence of periapical or periradicular radiolucency, a widened periodontal ligament space, physiological resorption, incomplete root formation, internal or external root resorption, pulp canal obliteration or pulp calcifications
* non-restorable tooth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Judd, DDS, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at The Hospital for Sick Children between September 2010 and September 2012.
Groups:
- MTA/FS Pulpotomy Group: Children randomized to this arm will undergo a mineral trioxide aggregate (MTA) pulpotomy after hemostasis is achieved using ferric sulfate (FS).
  Mineral trioxide aggregate/ferric sulfate (MTA/FS) pulpotomy: After complete removal of all caries, if a pulp exposure is detected the pulp chamber will be opened and vital coronal pulp to a depth of 2mm below free gingival margin will be removed. A solution of ferric sulfate will be applied to the amputated pulp surface and then flushed with water. MTA paste is then used to cover over the exposed amputated pulp surface.
- RCT Group: Children randomized to this group will undergo the root canal therapy (RCT) technique.
  Root canal therapy (RCT): After complete removal of all caries, if a pulp exposure is detected the pulp chamber will be opened and the pulp tissue removed. The canal will be irrigated with water and then filled with non-reinforced ZOE.
Period: Overall Study
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Started | 40 (100 incisors were treated in the MTA/FS pulpotomy group) | 30 (72 incisors were treated in the RCT group)
Completed | 40 (100 incisors were treated in the MTA/FS pulpotomy group) | 30 (72 incisors were treated in the RCT group)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The MTA/FS group consisted of 100 incisors in 40 subjects (19 males; 21 females) and the RCT group consisted of 72 primary incisors in 30 subjects (14 males; 16 females).
Groups:
- Total: Total of all reporting groups
Arm/Group | MTA/FS Pulpotomy Group | RCT Group | Total
Number analyzed (Participants) | 40 | 30 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 30 | 70
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 19 | 14 | 33
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 30 | 70
Incisors [Number; unit: incisors] | 100 | 72 | 172

OUTCOME MEASURES:

1. Primary Outcome: Comparison of MTA/FS Pulpotomy Versus RCT Treated Incisors With Acceptable Radiographic Outcome at 12 Months Post-procedure.
Description: Two disinterested pediatric dentists classified each treated incisor into one of three outcomes: N=incisor without pathologic change; Po=pathologic change present, follow-up recommended; and Px=pathologic change present, extract. Incisors rated N or Po were considered an acceptable radiographic outcome while incisors rated as Px were considered unacceptable.
Time Frame: 12 months after the procedure
Measure: Number; unit: Proportion of incisors
Units Other Than Participants: Incisors
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Number analyzed (Participants) | 40 | 30
Number analyzed (Incisors) | 100 | 72
Proportion of incisors | .97 | .92
Statistical Analysis 1: Comparison: MTA/FS Pulpotomy Group vs RCT Group; Radiographic outcomes were compared using univariate repeated measures logistic regression. A binary logistic generalized estimating equation model was used to analyze predictor variables such as age, gender, tooth and treatment provider between the treatment groups; Test type: Superiority or Other; p = .15, Chi-squared; Odds Ratio (OR) = .34, 95% CI 2-sided [.08 to 1.49]

2. Primary Outcome: Comparison of MTA/FS Pulpotomy Versus RCT Treated Incisors With Acceptable Radiographic Outcomes 18 Months Post-procedure.
Description: as for outcome 1
Time Frame: 18 months after the procedure
Measure: Number; unit: Proportion of incisors
Units Other Than Participants: Incisors
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Number analyzed (Participants) | 40 | 30
Number analyzed (Incisors) | 100 | 72
Proportion of incisors | .93 | .92
Statistical Analysis 1: Comparison: MTA/FS Pulpotomy Group vs RCT Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .38, Chi-squared; Odds Ratio (OR) = .6, 95% CI 2-sided [.19 to 1.89]

3. Secondary Outcome: Comparison of MTA/FS Pulpotomy Versus RCT Treated Incisors With Unacceptable Clinical Outcome at 12 Months Post-procedure.
Description: Pulp treated incisors presenting with spontaneous pain, tenderness to percussion, fistula/sinus tract, soft tissue swelling and/or pathological tooth mobility were considered unacceptable clinical outcomes. Clinical outcomes between the MTA/FS pulpotomy and RCT groups were compared using Fisher's Exact test.
Time Frame: 12 months after the procedure
Measure: Number; unit: Proportion of incisors
Units Other Than Participants: Incisors
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Number analyzed (Participants) | 40 | 30
Number analyzed (Incisors) | 100 | 72
Proportion of incisors | .98 | 1.0
Statistical Analysis 1: Comparison: MTA/FS Pulpotomy Group vs RCT Group; A binary logistic generalized estimating equation (GEE) model was used to analyze predictor variables such as age, gender, tooth and treatment provider between the treatment groups for radiographic and clinical outcomes; Test type: Superiority or Other; p = .51, Fisher Exact

4. Secondary Outcome: Comparison of MTA/FS Pulpotomy Versus RCT Treated Incisors With Unacceptable Clinical Outcome at 18 Months Post-procedure.
Description: Pulp treated incisors presenting with spontaneous pain, tenderness to percussion, fistula/sinus tract, soft tissue swelling and/or pathological tooth mobility were considered unacceptable clinical outcomes.
Time Frame: 18 months after the procedure
Measure: Number; unit: Proportion of incisors
Units Other Than Participants: Incisors
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Number analyzed (Participants) | 40 | 30
Number analyzed (Incisors) | 100 | 72
Proportion of incisors | .97 | .98
Statistical Analysis 1: Comparison: MTA/FS Pulpotomy Group vs RCT Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = .64, Fisher Exact

5. Secondary Outcome: MTA/FS Pulpotomy and RCT Treated Incisor Survival
Description: Kaplan-Meier survival curves were generated for the MTA/FS pulpotomy and RCT treatment groups. One treated incisor was selected by random draw from each subject for survival analysis to preserve independence of observations. The log-rank test was used to statistically compare survival of incisors.
Time Frame: 12 and 18 months
Population: Four participants in the MTA/FS and two participants in the RCT group did not have data collected due to lost to follow-up. Remaining participants were censored if lost to follow-up, exfoliated, lost to trauma or had a non-occurrence of a failure before the trial end.
Measure: Number; unit: Proportion of participants
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Number analyzed (Participants) | 36 | 28
Proportion of participants
  Survival at 12 months | 1 | .97
  Survival at 18 months | .94 | .97
Statistical Analysis 1: Comparison: MTA/FS Pulpotomy Group vs RCT Group; Test type: Superiority or Other; p = .11, Log Rank — The p-value represents the survival rate from the Kaplan-Meier survival analysis from 6 to 36 months

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | MTA/FS Pulpotomy Group | RCT Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/30
Other Adverse Events (participants affected / at risk) | 0/40 | 0/30

LIMITATIONS AND CAVEATS:
Limitations of the study design included no blinding of personnel providing treatment or raters assessing clinical and radiographic outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No